CLINICAL TRIAL: NCT01676961
Title: Phase II Trial Evaluating the Efficacy and Safety of Romiplostim (Nplate) Treatment of Chemotherapy Induced Thrombocytopenia in Patients With Multiple Myeloma
Brief Title: Romiplostim in Increasing Low Platelet Counts in Patients With Multiple Myeloma Receiving Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left the institution
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 10-02429; P30CA016087 (NIH)
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Results first posted 2017-09-05 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-09

CONDITIONS: Refractory Multiple Myeloma; Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma; Thrombocytopenia
MeSH Terms: conditions — Multiple Myeloma; Thrombocytopenia | interventions — romiplostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Supportive care (romiplostim) (Experimental): Patients receive romiplostim SC once weekly for up to 6 weeks. Patients achieving a platelet count > 50 x 10^9 then receive romiplostim once weekly during 1 course of chemotherapy and may continue for as long as benefit is seen..
  Interventions: Biological: romiplostim

INTERVENTIONS:
Biological: romiplostim — Given SC
  Other Names: AMG 531; Amgen megakaryopoiesis protein 2; Nplate

SUMMARY:
This phase II trial studies how well romiplostim works in increasing low platelet counts in patients with multiple myeloma receiving chemotherapy. Romiplostim may cause the body to make platelets after chemotherapy

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if Nplate (romiplostim) is capable of increasing platelet counts to > 50 x 10^9/L for greater than 2 weeks in myeloma patients with chemotherapy induced thrombocytopenia.

SECONDARY OBJECTIVES:

I. To evaluate the toxicity of romiplostim in this patient population by standard Common Toxicity Criteria (CTC).

II. To determine any increase in thrombosis or marrow fibrosis.

OUTLINE:

Patients receive romiplostim subcutaneously (SC) once weekly for up to 6 weeks. Patients achieving a platelet count > 50 x 10^9 then receive romiplostim once weekly during 1 course of chemotherapy and may continue for as long as benefit is seen.

After completion of study treatment, patients are followed up every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Subject is not pregnant or breast feeding, and cannot become pregnant within 30 days after the end of treatment
* Female subject of child bearing potential must be willing to use, in combination with her partner, 2 forms highly effective contraception during treatment and for 1 month after the end of treatment
* Diagnosis of any stage of multiple myeloma based on standard criteria as follows:

  * Major criteria

    1. Plasmacytomas on tissue biopsy
    2. Bone marrow plasmacytosis (> 30% plasma cells)
    3. Monoclonal immunoglobulin spike on serum electrophoresis (immunoglobin G [IgG] > 3.5 G/dL or immunoglobin A [IgA] > 2.0 G/dL) or kappa or lambda light chain excretion > 1 G/day on 24 hour urine protein electrophoresis
  * Minor criteria

    1. Bone marrow plasmacytosis (10 to 30% plasma cells)
    2. Monoclonal immunoglobulin present but of lesser magnitude than given under major criteria
    3. Lytic bone lesions
    4. Normal immunoglobin M (IgM) < 50 mg/dL, IgA < 100 mg/dL, or IgG < 600 mg/dL
  * Any of the following sets of criteria will confirm the diagnosis of multiple myeloma:

    * Any two of the major criteria
    * Major criterion 1 plus minor criterion b, c, or d
    * Major criterion 3 plus minor criterion a or c
    * Minor criteria a, b and c or a, b and d
* Karnofsky performance status >= 50
* Platelet count =< 50 x 10^9/L untransfused of at least 2 weeks duration, secondary to prior chemotherapy. If there is a platelet count of > or = 50 x 10(9)/L after a transfusion, that value will be discounted.

This may include a combination regimen including lenalidomide; these regimens will include dexamethasone, cyclophosphamide, etoposide, cisplatin (DCEP), Velcade with Doxil, Cytoxan and/or lenalidomide; patients who have thrombocytopenia (CIT) from lenalidomide or from radiation therapy alone will not be allowed

* Calculated or measured creatinine clearance >= 30 mL/min

Exclusion Criteria:

* POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein [M-protein] and skin changes)
* Plasma cell leukemia
* Receiving steroids daily for other medical conditions, e.g., asthma, systemic lupus erythematosus, rheumatoid arthritis
* Infection not controlled by antibiotics
* Human immunodeficiency virus (HIV) infection; patients should provide consent for HIV testing according to the institution's standard practice
* Known active hepatitis B or C
* Patient had myocardial infarction within 6 months prior to enrollment, New York Hospital Association (NYHA) class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities; prior to study entry, any electrocardiogram (ECG) abnormality at screening must be documented by the investigator as not medically relevant
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy
* Other serious medical or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol
* Female subject is pregnant or lactating; confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (hCG) pregnancy test result obtained during screening; pregnancy testing is not required for postmenopausal or surgically sterilized women
* Patient has > 1.5 x upper limit of normal (ULN) total bilirubin
* Patients with existing deep venous thrombosis will be excluded
* Patients receiving maintenance therapy with myelosuppressive medications such as lenalidomide will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amitabha Mazumder, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Cancer Institute, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Supportive Care (Romiplostim)
Started | 5
Completed | 0
Not Completed | 5
Not completed — Death | 3
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Confirmed diagnosis of multiple myeloma.
Arm/Group | Supportive Care (Romiplostim)
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Have Responded
Description: Response is defined as platelet increases to greater than 50 x 10^9/L for more than 2 weeks.
Time Frame: 8 weeks
Population: Data was not analyzed. Dr. Mazumder left institution and data was not analyzed.
Arm/Group | Supportive Care (Romiplostim)
Number analyzed (Participants) | 0

2. Secondary Outcome: Percentage of Patients Who Experienced Thrombosis or Marrow Fibrosis
Time Frame: Up to 1.5 years
Population: Patient data was not analyzefd
Arm/Group | Supportive Care (Romiplostim)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 4 Months
Arm/Group | Supportive Care (Romiplostim)
All-Cause Mortality (participants affected / at risk) | 4/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No